CLINICAL TRIAL: NCT00691912
Title: Extended Dose Frequency 1st-line Therapy of Metastatic Breast Cancer With Paclitaxel and Liposomal Doxorubicin (Myocet®)
Brief Title: Therapy of Metastatic Breast Cancer With Paclitaxel and Liposomal Doxorubicin
Acronym: MyoPac
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due because recrutation.was much slower as anticipated.
Sponsor: Claudia Lorenz-Schlüter (Other)
Responsible Party: Sponsor-Investigator, Claudia Lorenz-Schlüter, member of CRO, University of Magdeburg
Organization: University of Magdeburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4102000
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocet/Paclitaxel (Experimental): 20 mg/m² Myocet® as 30-minutes infusion on day 1,8,15 80 mg/m² Paclitaxel as 60-minutes infusion on day 1,8,15 q21d
  Interventions: Drug: liposomal Doxorubicin; Drug: Myocet / Paclitaxel

INTERVENTIONS:
Drug: liposomal Doxorubicin — 20 mg/m² Myocet® as 30-minutes infusion on day 1,8,15 80 mg/m² Paclitaxel as 60-minutes infusion on day 1,8,15 q21d
  Other Names: Myocet
Drug: Myocet / Paclitaxel — 20 mg/m² Myocet® as 30-minutes infusion on day 1,8,15 80 mg/m² Paclitaxel as 60-minutes infusion on day 1,8,15 q21d

SUMMARY:
Today metastatic breast cancer is regarded as cureless. The treatment is palliative in intent and the goals of treatment include improvement of quality of life and if possible prolongation of life. Treatment in metastatic cancer will usually involve hormone therapy and/or chemotherapy. Weekly application of chemotherapeutical drugs may lead to less drug concentrations in healthy tissue and therefore toxicities maý be reduced.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy of females. In Germany about 46,000 women come down with breast cancer yearly.

Present therapies cannot cure the metastatic disease, the main focus is improvement of quality of life and prolongation of life. It is therefore necessary to test new substances and/or new combinations and therapy concepts. Among the most active cytotoxic agents used in advanced breast cancer are the anthracyclines. Since conventional anthracyclines are often used as adjuvant or neoadjuvant therapy their cardiotoxicity restricts their use in the therapy of the advanced disease.

Liposomal encapsulated doxorubicin shows better activity than conventional doxorubicin combined with reduced cardiotoxicity.

Weekly applied cytotoxic agents show a better toxicity profile and hence the cumulative dosis can be increased. It is expected that the combination of liposomal encapsulated doxorubicin with paclitaxel given weekly shows improved results in the therapy of metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women >/= 18 years with histologically proven metastatic breast cancer
* No prior chemotherapy in the advanced situation
* ECOG </= 2
* Adequate bone marrow reserve
* left ventricular ejection fraction (LVEF) >/= 50, measured within 4 weeks before study treatment
* Existence of written informed consent

Exclusion Criteria:

* Previous high dose therapy with stem cell support
* Prior adjuvant treatment with cumulative anthracycline dose of 600 mg/m² Epirubicin, 300 mg/m² Doxorubicin, 80 mg/m² Mitoxantrone
* Concomitant hormon- or chemotherapy or radiation therapy
* Her2/neu overexpression
* pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
progression free survival assessed by imaging procedures | after 6 weeks, 12 weeks, 18 weeks

SECONDARY OUTCOMES:
toxicity, quality of life | every 3 weeks
response rate, overall survival | 28 d after last Chemotherapy, up then every 3 months for 1 and a half year, and up then every 6 months until 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Bischoff, Dr. med., Principal Investigator — Klinikum der Otto-von-Guericke Universität Magdeburg, Frauenklinik
Locations (1):
- Klinikum der Otto-von Guericke Universität Magdeburg, Frauenklinik, Magdeburg, Saxony-Anhalt, Germany